CLINICAL TRIAL: NCT00005887
Title: A Phase III, Randomized, Open-Label, Comparative Study of Standard Whole Brain Radiation Therapy With or Without RSR13 in Patients With Brain Metastases
Brief Title: Radiation Therapy With or Without RSR13 in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067957; ALLOS-RSR13RT-009
Record Dates: First submitted 2000-06-02; First posted 2003-08-29 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — efaproxiral; Radiotherapy

INTERVENTIONS:
Drug: efaproxiral
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as RSR13 may make tumor cells more sensitive to radiation therapy.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy to the brain with or without RSR13 in treating patients who have brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the median survival time in patients with brain metastases after receiving treatment with whole brain radiotherapy with or without RSR13.
* Compare the response rate to these treatment regimens in these patients.
* Compare the time to progression after receiving these treatment regimens in these patients.
* Compare quality of life in these patients receiving these treatment regimens.
* Compare cause of death (neurologic vs nonneurologic death) in these patients after receiving these treatment regimens.
* Determine the safety of RSR13 in these patients.
* Assess the pharmacokinetics of RSR13 in these patients.

OUTLINE: This is a randomized, open label, comparative, multicenter study. Patients are stratified according to the Radiation Therapy Oncology Group RPA Class (I vs II). Patients are further stratified within the RPA class II stratum according to site of primary cancer (non-small cell lung cancer vs breast vs other). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive whole brain radiotherapy 5 days a week for two weeks in conjunction with supplemental oxygen breathing.
* Arm II: Patients receive RSR13 IV over 30 minutes followed by whole brain radiotherapy and supplemental oxygen breathing as in arm I.

Quality of life is assessed at the first and last day of radiotherapy, at 1 month, 3 months, and then every 3 months until disease progression.

Patients are followed at 1 month, 3 months, every 3 months until disease progression, and then for survival.

PROJECTED ACCRUAL: A maximum of 408 (204 per treatment arm) patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiographically, histologically, or cytologically confirmed brain metastases with histologically or cytologically confirmed primary malignancy except the following:

  * Small cell lung cancer, germ cell tumors, and lymphomas
* No leptomeningeal metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 10 g/dL
* WBC at least 2,000/mm3
* Platelet count at least 75,000/mm3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT and AST no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Pulmonary:

* Forced vital capacity and forced expiratory volume at least 50% of normal in patients with significant intrathoracic tumor involvement, chronic obstructive pulmonary disease, interstitial lung disease, or pulmonary embolism
* Resting and exercise oxygen saturation at least 90% on room air

Other:

* No other concurrent active malignancy from a second histologic site
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy or immunotherapy for brain metastases
* At least 28 days since prior investigational biologic therapy

Chemotherapy:

* No prior chemotherapy for brain metastases
* No chemotherapy for brain metastases for at least one month following radiation therapy
* At least 7 days since prior chemotherapy for primary tumor or extracranial metastases
* No planned chemotherapy during radiation therapy

Endocrine therapy:

* No prior hormonal therapy for brain metastases
* Prior or concurrent corticosteroid therapy allowed

Radiotherapy:

* No prior whole brain radiotherapy for brain metastases
* No prior stereotactic radiosurgery for brain metastases

Surgery:

* Prior surgery allowed for brain metastases if at least one measurable lesion remains

Other:

* At least 28 days since prior investigational drug or device
* No prior RSR13

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02 (Actual); Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences
Locations (73):
- United States (35):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - California Cancer Care, Inc., Greenbrae, California
  - Scripps Green Hospital & Scripps Clinic, La Jolla, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - Citrus Memorial Hospital, Inverness, Florida
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Ochsner Clinic, New Orleans, Louisiana
  - Harbor Hospital Center, Baltimore, Maryland
  - St. Agnes Healthcare, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - East Coast Radiation Oncology, Toms River, New Jersey
  - Millard Fillmore Hospital, Buffalo, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Memphis Regional Brain Tumor Center, Memphis, Tennessee
  - Boston Baskin Cancer Group, University Tennessee Oncology/Hematology Group, Memphis, Tennessee
  - U.S. Oncology Research Inc., Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Center for Radiation Oncology, Danville, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Australia (4):
  - Royal Prince Alfred Hospital Medical Center, Sydney, New South Wales
  - Queensland Radium Institute, Herston, Queensland
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Austin and Repatriation Medical Centre, Heidelberg West, Victoria
- Belgium (4):
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels (Bruxelles)
  - UZ De Pintelaan, Ghent
  - U.Z. Gasthuisberg, Leuven
- Canada (15):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- France (4):
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - CHU de la Timone, Marseille
  - Hopital de Montbeliard, Montbéliard
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (2):
  - Radiologische Uniklink, Freiburg im Breisgau
  - Universitats-Krankenhaus Eppendorf, Hamburg
- Hungary (5):
  - Uzsoki Hospital, Budapest
  - University of Debrecen, Debrecen
  - Petz Aladar County Hospital, Gydr
  - Borsod-Abauj-Zemplen County Hospital, Miskolc
  - Szeged University, Szeged
- Italy (2):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Istituto Europeo Di Oncologia, Milan
- United Kingdom (2):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Western General Hospital, Edinburgh, Scotland

REFERENCES:
- [Result] Suh JH, Stea B, Nabid A, Kresl JJ, Fortin A, Mercier JP, Senzer N, Chang EL, Boyd AP, Cagnoni PJ, Shaw E. Phase III study of efaproxiral as an adjunct to whole-brain radiation therapy for brain metastases. J Clin Oncol. 2006 Jan 1;24(1):106-14. doi: 10.1200/JCO.2004.00.1768. Epub 2005 Nov 28. PMID 16314619
- [Result] Nabid A, Kresl J, Stea B, et al.: Standard whole brain radiation (WBRT) with supplemental oxygen (O2) with or without RSR13 (efaproxiral) in patients with brain metastases originating from NSCLC: results of a subgroup analysis. [Abstract] J Clin Oncol 22 (Suppl 14): A-7115, 645s, 2004.
- [Result] Shaw E, Stea B, Pinter T, et al.: Pharmacokinetics (PK) of RSR13 (efaproxiral) predict survival in patients with brain metastases randomized to receive whole brain radiation therapy (WBRT) with or without RSR13 (REACH RT-009). [Abstract] J Clin Oncol 22 (Suppl 14): A-1561, 122s, 2004.
- [Result] Stea B, Suh J, Shaw E, et al.: Efaproxiral (EFAPROXYN) as an adjunct to whole brain radiation therapy for the treatment of brain metastases originating from breast cancer: updated survival results of the randomized REACH (RT-009) study. [Abstract] Breast Cancer Res Treat 88 (1): A-4064, 2004.
- [Result] Suh J, Stea BD, Nabid A, et al.: Prognostic factors for survival in patients with brain metastases enrolled on a worldwide phase 3 randomized trial of 538 patients (study RSR13 RT-009). [Abstract] Int J Radiat Oncol Biol Phys 60 (1 Suppl 1): A-60, S165, 2004.
- [Result] Suh J, Stea B, Nabid A, et al.: Standard whole brain radiation therapy (WBRT) with supplemental oxygen (O2), with or without RSR13 (efaproxiral) in patients with brain metastases: results of the randomized REACH (RT-009) study. [Abstract] J Clin Oncol 22 (Suppl 14): A-1534, 115s, 2004.